CLINICAL TRIAL: NCT06112327
Title: Long-term Follow-up Study of Investigational Gene-editing Therapies in Participants with or At High Risk for Cardiovascular Disease
Brief Title: Long-term Follow-up of Participants Dosed with an Investigational Gene Editing Therapy for Cardiovascular Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Verve Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LTF-001
Record Dates: First submitted 2023-10-12; First posted 2023-11-01 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Atherosclerotic Cardiovascular Disease; Heterozygous Familial Hypercholesterolemia; Hypercholesterolemia
Keywords: LTF-001; Cardiovascular Disease; Gene Editing; Familial Hypercholesterolemia; Base Editing
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Cardiovascular Diseases; Hyperlipoproteinemia Type II

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
LTF-001 is a long-term follow-up study of participants who received an investigational gene-editing therapy developed by the sponsor to evaluate the long-term effects of the investigational therapy. Participants will be followed for a total of 15 years after the first administration of the gene-editing therapy.

ELIGIBILITY:
Inclusion Criteria

1. A participant has completed or discontinued from a Verve sponsored clinical study in which they received at least one dose of study drug.
2. A participant has provided informed consent for LTF-001.

Exclusion Criteria: N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who received an investigational gene-editing therapy developed by the sponsor.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-06-09 (Actual); Primary Completion 2039-10 (Estimated); Study Completion 2039-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-related adverse events (AEs), serious adverse events (SAEs) and other events of interest using CTCAE 5.0 to assess the long-term safety of gene-editing therapies. | up to 15 years
  To assess the long-term safety of gene-editing therapies, the following will be assessed:
  Incidence of treatment-related adverse events (AEs), serious adverse events (SAEs) and any CTCAE grade 3 or higher AEs.

SECONDARY OUTCOMES:
Percent and absolute change from baseline of lipid concentrations over time after administration of a gene-editing therapy. | up to 15 years
  Blood samples will be collected to assess percent change from baseline in lipid concentrations (including LDL-C).
Percent and absolute change from baseline of target biomarkers over time after administration of a gene-editing therapy. | up to 15 years
  Blood samples will be collected to assess percent change from baseline in target biomarkers.

CONTACTS AND LOCATIONS:
Locations (3):
- New Zealand (2):
  - Clinical Study Center, Auckland
  - Clinical Study Center, Christchurch
- Clinical Study Center, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No